CLINICAL TRIAL: NCT00002715
Title: A Phase II Pilot Study of Short Term (12 Week) Combination Chemotherapy (Stanford V) in Unfavorable Hodgkin's Disease
Brief Title: Combination Chemotherapy in Treating Patients With Advanced Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-13467; SUMC-G2/G3 (Other: Stanford University Medical Center); CDR0000064551 (Other: Stanford University Medical Center); SQL 76234 (Other: Stanford University Medical Center); NCI-H96-0806 (Other: Old NCI)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Lymphoma
Keywords: Stage I adult Hodgkin lymphoma; Stage II adult Hodgkin lymphoma; Stage III adult Hodgkin lymphoma; Stage IV adult Hodgkin lymphoma; Adult lymphocyte predominant Hodgkin lymphoma; Adult lymphocyte depletion Hodgkin lymphoma; Adult nodular sclerosis Hodgkin lymphoma; Adult mixed cellularity Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Bleomycin; Doxorubicin; Etoposide; Mechlorethamine; Prednisone; Vinblastine; Vincristine

ARMS (1):
- Combination Chemotherapy (Stanford V) (Experimental): A combination chemotherapy regimen consisting of mechlorethamine, doxorubicin hydrochloride, vinblastine, vincristine, bleomycin, etoposide and prednisone, administered on a compressed schedule
  Interventions: Biological: Bleomycin sulfate; Drug: Stanford V regimen; Drug: Doxorubicin hydrochloride; Drug: Etoposide; Drug: Mechlorethamine hydrochloride; Drug: Prednisone; Drug: Vinblastine; Drug: Vincristine sulfate

INTERVENTIONS:
Biological: Bleomycin sulfate — A component of the Stanford V regimen.
Drug: Stanford V regimen
Drug: Doxorubicin hydrochloride — A component of the Stanford V regimen.
Drug: Etoposide — A component of the Stanford V regimen.
Drug: Mechlorethamine hydrochloride — A component of the Stanford V regimen.
Drug: Prednisone — A component of the Stanford V regimen.
Drug: Vinblastine — A component of the Stanford V regimen.
Drug: Vincristine sulfate — A component of the Stanford V regimen.

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy in treating patients who have advanced Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of short term chemotherapy with the Stanford V regimen (mechlorethamine, doxorubicin, vinblastine, prednisone, vincristine, bleomycin, and etoposide) followed by, as indicated, consolidative radiotherapy in patients with stage IIB, IIIA, IIIB, or IV Hodgkin's lymphoma.
* Determine the initial response to 8 weeks of Stanford V chemotherapy in these patients.
* Assess the complete and partial response rate to 12 weeks of Stanford V chemotherapy in these patients.
* Determine the acute toxicity associated with this treatment.
* Determine the disease free interval and survival following Stanford V chemotherapy with or without consolidative radiotherapy in these patients.

OUTLINE: All patients are treated on Regimen A with the Stanford V Regimen; those with initial bulky, residual, or splenic disease who achieve a CR/PR proceed to Regimen B.

* Regimen A: Patients receive mechlorethamine IV on weeks 1, 5, and 9; doxorubicin and vinblastine IV on weeks 1, 3, 5, 7, 9, and 11; vincristine and bleomycin IV on weeks 2, 4, 6, 8, 10, and 12; etoposide IV over 30-45 minutes for 2 consecutive days on weeks 3, 7, and 11; and prednisone orally every other day on days 1-84. Treatment continues for 8-12 weeks, depending on response, in the absence of disease progression or unacceptable toxicity.
* Regimen B: Patients begin radiotherapy 2-4 weeks after completion of Regimen A. Patients receive radiotherapy to lungs, pleura, and other extralymphatic sites for approximately 5 weeks.

Patients are followed for survival.

PROJECTED ACCRUAL: A total of 50 patients will be entered if at least 16 of the first 22 patients respond. As of 03/96, it is expected that a total of 45 patients each with stage III/IV disease and 40 with unfavorable stage II disease will be accrued.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed Hodgkin's lymphoma of any histology
* Unfavorable disease required

  * Clinical stage IIIA, IIIB, IV, or IIB (non-bulky)
  * Locally extensive stage I or II with either of the following:

    * Mediastinal mass greater than 1/3 the maximum intrathoracic diameter
    * Two or more extranodal sites

PATIENT CHARACTERISTICS:

Age:

* 18 to 60

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No prior malignancy except nonmelanomatous skin cancer
* No significant concurrent illness that precludes protocol participation

PRIOR CONCURRENT THERAPY:

* No prior treatment for Hodgkin's lymphoma

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 1989-04 (Actual); Primary Completion 2007-01 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra J. Horning, MD, Study Chair — Stanford University
Locations (1):
- Stanford Cancer Center at Stanford University Medical Center, Stanford, California, United States

REFERENCES:
- [Result] Horning SJ, Rosenberg SA, Hoppe RT. Brief chemotherapy (Stanford V) and adjuvant radiotherapy for bulky or advanced Hodgkin's disease: an update. Ann Oncol. 1996;7 Suppl 4:105-8. doi: 10.1093/annonc/7.suppl_4.s105. PMID 8836420
- [Result] Bartlett NL, Rosenberg SA, Hoppe RT, Hancock SL, Horning SJ. Brief chemotherapy, Stanford V, and adjuvant radiotherapy for bulky or advanced-stage Hodgkin's disease: a preliminary report. J Clin Oncol. 1995 May;13(5):1080-8. doi: 10.1200/JCO.1995.13.5.1080. PMID 7537796